CLINICAL TRIAL: NCT02254668
Title: Intracoronary Analysis of Cardiac Allograft Vasculopathy in Comparison to Coronary Artery Disease by Means of Optical Coherence Tomography
Brief Title: Intracoronary Analysis of Cardiac Allograft Vasculopathy by Means of Optical Coherence Tomography
Acronym: OCTandCAV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH_Nr. 2012-0409
Record Dates: First submitted 2013-12-29; First posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Intimal Proliferation; Immunosuppression
Keywords: intima; thickness; transplantation; cardiology; immunosuppression
MeSH Terms: interventions — Clinical Protocols; Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Certican®) (Experimental): Electronic (computer-assisted) randomization of an immunosuppressive protocol WITH Everolimus (Certican®). No protocol with Mycophenolate mofetil (CellCept®). Daily dosage administered depending on blood concentration (control interval 6-12 months)
  Interventions: Other: Protocol with Everolimus (Certican®)
- Mycophenolate mofetil (CellCept®) (Active Comparator): Electronic (computer-assisted) randomization of an immunosuppressive protocol WITHOUT Everolimus (Certican®), instead administration of Mycophenolate mofetil (CellCept®). No protocol with Everolimus (Certican®). Daily dosage administered depending on blood concentration (control interval 6-12 months)
  Interventions: Other: Protocol with Mycophenolate mofetil (CellCept®)

INTERVENTIONS:
Other: Protocol with Everolimus (Certican®) — Electronic (computer-assisted) randomization of an immunosuppressive protocol WITH Everolimus (Certican®).
  Other Names: Randomizaiton by SecuTrial
  Arms: Everolimus (Certican®)
Other: Protocol with Mycophenolate mofetil (CellCept®) — Electronic (computer-assisted) randomization of an immunosuppressive protocol WITHOUT Everolimus (Certican®), instead administration of Mycophenolate mofetil (CellCept®).
  Other Names: Randomizaiton by SecuTrial
  Arms: Mycophenolate mofetil (CellCept®)

SUMMARY:
Randomized prospective multi-center imaging study which investigates the impact of different immunosuppressive protocols (Everolimus (Certican®) or Mycophenolate mofetil (CellCept®)) on cardiac allograft vasculopathy (CAV) in heart transplanted patients. Maximal intima-thickness will be visualized by optical coherence tomography (OCT) to assess the progression of CAV.

DETAILED DESCRIPTION:
In summary, the aim of the study is to examine the effect of the immunosuppressive agent Everolimus (Certican) on the development of cardiac allograft vasculopathy (CAV).

Therefore the study is divided in three sections:

Substudy 1: Evaluation of morphological differences between between CAD and CAV.

Substudy 2: Analysis of cardiovascular risk factors (e.g. hypertension) under a specific immunosuppressive protocol in patients with CAV.

Substudy 3: Prospective, randomized analysis of the influence of different immunosuppressive protocols in patients with CAV.

Primary endpoint of the study will be the adaption of intimal thickness after 10 years, analysed by means of optical coherence tomography.

In addition to the explanations above the most important in- and exclusion criteria are listed below:

Inclusion Criteria:

* Patients after heart transplantation
* Patients with coronary artery disease (CAD)
* Age 18-80 years

Exclusion Criteria:

* Contraindication of Everolimus/Sirolimus or adjuvants
* Renal insufficiency (Creatinine > 265 µmol/l)
* Cardiogenic shock or patients with Killip*-Class III or IV (*name)
* Pregnant or breast feeding females
* insufficient contraception (only for substudy 3)

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart transplantation
* Patient with coronary artery disease
* Age between 18 and 80 years

Exclusion Criteria:

* Renal insufficiency (> 265 µmol/l)
* Incapability to give informed consent
* Cardiogenic shock of patient with KILLIP III or IV
* pregnant or breast feeding females
* insufficient contraception (only for substudy 3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Intimal Thickness | Assessment intervals of patients with CAV is 1 year and 2 years in patients without CAV
  Assessment is usually performed by intracoronary angiography and endomyocardial biopsy which is routinely performed <1 year after heart transplantation. Furthermore, assessment interval will be defined according to the result of these investigational procedures. If there is a diagnosis of CAV the interval will be one year, if not a follow-up examination in two years will be sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Templin, MD, PhD, Principal Investigator — University Hospital Zurich (Switzerland), Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- See also: Informations about Optical Coherence Tomography (OCT) — http://www.octnews.org